CLINICAL TRIAL: NCT01506180
Title: In-Hospital Comprehensive Geriatric Assessment in Aged Acute Medical Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Merete Gregersen, Principal Investigator, Master of Health Science, University of Aarhus
Other Study IDs: CGA-GD-2011
Record Dates: First submitted 2011-11-02; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Acute Disease
Keywords: acute medical care; comprehensive geriatric assessment; Health Services for the Aged; Geriatric Assessment; Geriatrics; Aged
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients admitted to Geriatric Department: The patients receive comprehensive geriatric assessment
- Patients admitted to general medical departments: This group do not receive comprehensive geriatric assessment

SUMMARY:
The purpose of this study is to compare acute ill elderly medical patients in a geriatric department with general medical departments, and to examine the effects of comprehensive geriatric assessment in the geriatric setting compared with general medical care.

DETAILED DESCRIPTION:
Design:

1) a cross-sectional study followed by 2) a subgroup study by retrospective follow-up

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the departments of medicine at Aarhus University Hospital either through the emergency medical ward or directly to the medical wards in the period from January 1, 2009 to December 31, 2010.

Exclusion Criteria:

* patients admitted to the neurology-, cardiology-, nephrology- or haematology departments, and patients discharged directly to their homes from the emergency medical ward.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Acute medical patients aged 80 years or older
Sampling Method: Probability Sample
Enrollment: 3877 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Comorbidity | At hospital admission (day 1)
  By Charlsons Comorbidity Index
Length of hospital stay | Number of days of hospitalization an expected average of 8 days
  Participants will be followed for the duration of hospital stay, an expected average of 8 days.

SECONDARY OUTCOMES:
Acute readmission | 30 days and 90 days
  The number of acute readmissions in the participants within 30 days and 90 days after the discharge, respectively.
Mortality | Within 30 days after hospital admission
  The number of short-term mortality in the participants within 30 days after hospital admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Gregersen M, Pedersen AB, Damsgaard EM. Comprehensive geriatric assessment increases 30-day survival in the aged acute medical inpatients. Dan Med J. 2012 Jun;59(6):A4442. PMID 22677240